CLINICAL TRIAL: NCT02639559
Title: A Phase II Study Evaluating the Safety and Efficacy of BL-8040 for the Mobilization of Donor Hematopoietic Stem Cells and Allogeneic Transplantation in Patients With Advanced Hematological Malignancies
Brief Title: Safety and Efficacy of BL-8040 for the Mobilization of Donor Hematopoietic Stem Cells and Allogeneic Transplantation in Patients With Advanced Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201602037
Record Dates: First submitted 2015-12-17; First posted 2015-12-24 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Non-Hodgkin's Lymphoma; Non-Hodgkin Lymphoma; Hodgkin Disease; Hodgkins Disease; Hodgkin's Disease; Multiple Myeloma; Myelodysplastic Syndrome; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — 4-fluorobenzoyl-TN-14003; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Donors (Experimental): -Donors will receive subcutaneous (SC) BL-8040 in the morning (Day 1) followed by leukapheresis approximately 180 minutes (up to 270 minutes) after the injection per institutional protocol. If the donor does not reach the collection goal for mobilization (≥ 5.0 x 10^6 CD34+ cells/kg), a second leukapheresis will be performed on Day 2 (24 hours ± 2 hours from the BL-8040 injection) in an effort to reach a total of ≥ 5 x 10^6 CD34+ cells/kg and at least ≥ 2 x 10^6 CD34+ cells/kg from the combined collections.
  Interventions: Drug: BL-8040; Procedure: Leukapheresis
- Arm 2: Recipients (Experimental): -All or part of the leukapheresis product will be infused into the recipient per institutional guidelines. The day of the infusion will be considered Day 0; if the infusion occurs over multiple days, the final day of infusion will be considered Day 0
  Interventions: Procedure: Hematopoietic cell transplant

INTERVENTIONS:
Drug: BL-8040
  Arms: Arm 1: Donors
Procedure: Leukapheresis
  Arms: Arm 1: Donors
Procedure: Hematopoietic cell transplant
  Arms: Arm 2: Recipients

SUMMARY:
Current protocols use G-CSF to mobilize hematopoietic progenitor cells from matched sibling and volunteer unrelated donors. Unfortunately, this process requires four to six days of G-CSF injection and can be associated with side effects, most notably bone pain and rarely splenic rupture. BL-8040 is given as a single SC injection, and collection of cells occurs on the same day as BL-8040 administration. This study will evaluate the safety and efficacy of this novel agent for hematopoietic progenitor cell mobilization and allogeneic transplantation based on the following hypotheses:

* Healthy HLA-matched donors receiving one injection of BL-8040 will mobilize sufficient CD34+ cells (at least 2.0 x 10^6 CD34+ cells/kg recipient weight) following no more than two leukapheresis collections to support a hematopoietic cell transplant.
* The hematopoietic cells mobilized by SC BL-8040 will be functional and will result in prompt and durable hematopoietic engraftment following transplantation into HLA-identical siblings with advanced hematological malignancies using various non-myeloablative and myeloablative conditioning regimens and regimens for routine GVHD prophylaxis.
* If these hypotheses 1 and 2 are confirmed after an interim safety analysis of the data, then the study will continue and include recruitment of haploidentical donors.

ELIGIBILITY:
Inclusion Criteria (DONOR):

* Age 18 to 70 years of age.
* ECOG performance status of 0 or 1.
* PART 1: Donor must be a 5/6 or 6/6 HLA-matched sibling willing to donate PBSC for transplant.
* PART 2: Donor must be a 5/6 or 6/6 HLA-matched sibling or 3/6 or 4/6 HLA haploidentical donor willing to donate PBSC for transplant. Haploidentical donors will be allowed to participate upon investigator decision and based on the data reached from 5/6 or 6/6 HLA matched transplant done during Part 1 of the study.
* Adequate organ function defined by:

  * serum creatinine within normal limits or a minimum creatinine clearance (CrCl) value of ≥ 60 ml/min calculated using the Modification of Diet in Renal Disease (MDRD) Study equation
  * AST, ALT and total bilirubin ≤ 2x institutional upper limit of normal.
* Women of childbearing potential and men must agree to use adequate contraception with two different forms, including one barrier method, during participation in the study and for 2 weeks following dosing with BL-8040. Abstinence is acceptable if this is the established and preferred contraception for the subject.
* Female subjects must have a negative urine or serum pregnancy test within 10 days prior to taking study medication if of childbearing potential or must be of non-childbearing potential. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the subject to be eligible. Non-childbearing potential is defined as:

  -≥ 45 years of age and has not had menses for > 2 years
* Amenorrheic for > 2 years without a hysterectomy and oophorectomy and a FSH value in the postmenopausal range upon pretrial (screening) evaluation
* Post-hysterectomy, oophorectomy, or tubal ligation.
* Able and willing to comply with the requirements of the protocol.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Inclusion Criteria (RECIPIENT):

* Age 18 to 75 years
* ECOG performance status of 0-2 (inclusive)
* One of the following diagnoses:

  * Acute myelogenous leukemia (AML) in 1st or subsequent remission
  * Acute lymphoblastic leukemia (ALL) in 1st or subsequent remission
  * Chronic myelogenous leukemia (CML) in chronic or accelerated phase
  * Non-Hodgkin lymphoma (NHL) or Hodgkin's disease (HD) in 2nd or greater complete remission, partial remission
  * Chronic lymphocytic leukemia (CLL)
  * Multiple myeloma (MM)
  * Myelodysplastic syndrome (MDS)
  * Myeloproliferative neoplasm (MPN) excluding primary or secondary myelofibrosis
* Adequate organ function defined by:

  * a creatinine clearance (CrCl) value of ≥ 60 ml/min by MDRD study equation
  * AST, ALT and a total bilirubin ≤ 2x institutional upper limit of normal.
* Adequate cardiac function with a left ventricular ejection fraction ≥ 40%.
* Adequate pulmonary function defined as NO severe or symptomatic restrictive or obstructive lung disease, and formal pulmonary function testing showing an FEV1 ≥50% of predicted and a DLCO ≥ 40% of predicted, corrected for hemoglobin.
* Female subjects must have a negative urine or serum pregnancy test if of childbearing potential or be of non-childbearing potential. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the subject to be eligible. Non-childbearing potential is defined as:

  *≥ 45 years of age and has not had menses for > 2 years
  * Amenorrheic for > 2 years without a hysterectomy and oophorectomy and a FSH value in the postmenopausal range upon pretrial (screening) evaluation
  * Post-hysterectomy, oophorectomy, or tubal ligation.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria (DONOR):

* Received any investigational agent within 30 days and/or 5 half-lives (of the other investigational agent), whichever is longer, of receiving BL-8040.
* Active HIV or hepatitis B or C infection
* Pregnant or breastfeeding.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known allergy or hypersensitivity to any of the test compounds, materials, or contraindication to test products.
* Any malignancies in the 2 years prior to baseline, excluding: basal cell carcinoma, in situ malignancy, low-risk prostate cancer, cervix cancer after curative therapy.
* A comorbid condition which, in the view of the investigators, renders the subject at high risk from treatment complications.

Exclusion Criteria (RECIPIENT):

* Recipient must not have received any investigational drug within 30 days of starting conditioning treatment.
* Pregnant or breastfeeding.
* Active HIV or hepatitis B or C infection.
* Any medical condition which, in the opinion of the clinical investigator, would interfere with the evaluation of the patient. Subjects with a clinically significant or unstable medical or surgical condition or any other condition that cannot be well-controlled by the allowed medications permitted in the study protocol that would preclude safe and complete study participation, as determined by medical history, physical examinations, ECG, laboratory tests, or chest-X-ray and according to the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2023-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Uy, M.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Northside Hospital Cancer Institute, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Started | 25 | 25
Completed | 24 | 22
Not Completed | 1 | 3
Not completed — Mobilization failure | 0 | 3
Not completed — Issues with vascular acess | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Donors | Arm 2: Recipients | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: years] | 55 [20 to 69] | 58 [26 to 71] | 55 [20 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 18 | 15 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 21 | 23 | 44
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 20 | 22 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Donors That Mobilize ≥ 2 x 10^6 CD34+ Cells/kg of Recipients Weight After a Single Injection of BL-8040 After no More Than Two Leukapheresis Collections (Arm 1 - Donors Only)
Time Frame: Up to Day 2
Population: This outcome measure is for Arm 1 - Donors only.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 24 | 0
Participants | 22 |

2. Secondary Outcome: Safety and Tolerability of BL-8040 in Healthy Donors as Measured by Number and Grade of Adverse Events (Arm 1 Donors Only)
Description: -Adverse events will be graded according to the NCI CTCAE version 4.03
Time Frame: Up to 5 years
Population: This outcome measure is for Donor Arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 25 | 0
Participants
  Grade 1/2 anemia | 17 |
  Grade 1/2 sinus bradycardia | 1 |
  Grade 1/2 sinus tachycardia | 2 |
  Grade 1/2 eye pain | 1 |
  Grade 1/2 watering eyes | 1 |
  Grade 1/2 nausea | 5 |
  Grade 1/2 oral dysesthesia | 6 |
  Grade 1/2 vomiting | 2 |
  Grade 1/2 chills | 1 |
  Grade 1/2 fatigue | 3 |
  Grade 1/2 fever | 1 |
  Grade 1/2 infusion related reaction | 1 |
  Grade 1/2 injection site reaction | 20 |
  Grade 1/2 localized edema | 1 |
  Grade 1/2 pain | 1 |
  Grade 1/2 vibration sensation | 1 |
  Grade 1/2 allergic reaction | 20 |
  Grade 1/2 papulopustular rash | 1 |
  Grade 1/2 bruising | 1 |
  Grade 1/2 hemoglobin increased | 1 |
  Grade 1/2 lymphocyte count decreased | 6 |
  Grade 3 lymphocyte count decreased | 1 |
  Grade 1/2 lymphocyte count increased | 22 |
  Grade 1/2 platelet count decreased | 22 |
  Grade 1/2 weight loss | 1 |
  Grade 1/2 white blood cell decreased | 2 |
  Grade 1/2 A1c increased | 1 |
  Grade 1/2 hyperglycemia | 2 |
  Grade 1/2 hyperkalemia | 1 |
  Grade 1/2 hypocalcemia | 10 |
  Grade 1/2 hypomagnesemia | 1 |
  Grade 1/2 arthralgia | 1 |
  Grade 1/2 bone pain | 2 |
  Grade 1/2 foot pain | 1 |
  Grade 1/2 numbness in arms | 1 |
  Grade 1/2 pain in extremity | 1 |
  Grade 1/2 dysesthesia | 1 |
  Grade 1/2 dizziness | 1 |
  Grade 1/2 dysgeusia | 1 |
  Grade 1/2 headache | 3 |
  Grade 1/2 paresthesia | 3 |
  Grade 1/2 insomnia | 1 |
  Grade 1/2 dyspnea | 1 |
  Grade 1/2 hypertension | 7 |
  Grade 3 hypertension | 4 |
  Grade 1/2 hypotension | 2 |

3. Secondary Outcome: Time to Neutrophil Engraftment Post-transplant in Patients Undergoing Allogeneic Stem Cell Transplant (Arm 2 Recipients Only)
Description: -Time to neutrophil engraftment is measured by determining the first of 3 consecutive measurements of neutrophil count ≥ 500/μL following conditioning regimen induced nadir.
Time Frame: Up to Day 28
Population: -Donors are not evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
days |  | 13 [11 to 26]

4. Secondary Outcome: Time to Platelet Engraftment Post-transplant in Patients Undergoing Allogeneic Stem Cell Transplant (Arm 2 Recipients Only)
Description: -Time to platelet engraftment is measured by determining the first of 3 consecutive measurements of platelet count ≥ 20,000/μL without platelet transfusion support for 7 days.
Time Frame: Through 90 days
Population: -Donors are not evaluable for this outcome measure. 1 recipient was not evaluable due to no platelet nadir and 1 recipient was not evaluable due to no engraftment.
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 20
days |  | 20 [15 to 41]

5. Secondary Outcome: Number of Recipients With Primary Graft Failure After Transplantation of Hematopoietic Cells Mobilized With BL-8040 (Arm 2 Recipients Only)
Time Frame: Up to 1 year after transplantation
Population: -Donors are not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
Participants |  | 0

6. Secondary Outcome: Incidence of Secondary Graft Failure After Transplantation of Hematopoietic Cells Mobilized With BL-8040 (Arm 2 Recipients Only)
Time Frame: Up to 1 year after transplantation
Population: -Donors are not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
Participants |  | 0

7. Secondary Outcome: Cumulative Incidence of Grade 2-4 Acute Graft Versus Host Disease (GvHD) as Measured by Minnesota Acute GVHD Criteria (Arm 2 Recipients Only)
Description: * Acute GVHD rate and worst severity is noted
  * 4 organ categories (skin, liver, lower GI, and upper GI)
  * Skin: Grade I: 1-2 , Grade II: 3, Grade III: N/A, Grade IV: 4
  * Liver: Grade I: 0, Grade II: 1, Grade III: 2-4, Grade IV: N/A
  * Lower GI: Grade I: 0, Grade II: 1: Grade II: 2-3: Grade IV: 4
  * Upper GI: Grade I: 0, Grade II: 1, Grade III: N/A, Grade IV: N/A
  * The cumulative incidence of grade 2-4 acute GVHD was determined using competing risk analysis. Competing risks for acute GVHD were death, relapse, and graft failure.
Time Frame: Day 100
Population: -Donors are not evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
proportion of participants |  | 0.3636 [0.1690 to 0.5623]

8. Secondary Outcome: Cumulative Incidence of Chronic GvHD in Patients Who Have Undergone Transplantation of Hematopoietic Cells Mobilized With BL-8040 (Arm 2 Recipients Only)
Description: * Chronic GVHD rate and severity for the first 365 days after PBSC infusion will be assessed based on the NIH criteria
  * The cumulative incidence of chronic GVHD was determined using competing risk analysis. Competing risks for acute GVHD were death, relapse, and graft failure.
Time Frame: From Day 100 through 1 year after transplantation
Population: -Donors are not evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
proportion of participants |  | 0.5000 [0.2676 to 0.6946]

9. Secondary Outcome: Number of Participants Who Collect 5 x 106 CD34+ Cells/kg of Recipient Weight in a Single Leukapheresis and in 2 Leukapheresis Sessions (Arm 1 Donors Only)
Time Frame: Up to Day 2
Population: -Recipients are not evaluable for this outcome measure. -Only donors who received 1.25 mg/kg of BL-8040 were evaluable for this outcome measure (the 1st 10 donors received 1.00 mg/kg of BL-8040)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 9 | 0
Participants | 9 |

10. Secondary Outcome: Incidence of CMV Reactivation After Transplantation of Hematopoietic Cells Mobilized With BL-8040 in CMV Seropositive Recipients
Description: -CMV reactivation will be defined as a positive test for CMV viremia as determined by an antigenemia assay or quantitative PCR that results in the administration of antiviral treatment directed against CMV
Time Frame: Up to 1 year after transplantation
Population: -Donors are not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
Participants |  | 8

11. Secondary Outcome: Cumulative Incidence of Treatment-related Mortality After Transplantation of Hematopoietic Cells Mobilized With BL-8040 (Arm 2 Recipients Only)
Description: -Death that results from a transplant procedure related complication (e.g. infection, organ failure, hemorrhage, GVHD) rather than from relapse of the underlying disease or an unrelated cause
Time Frame: Up to 1 year after transplantation
Population: -Donors are not evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
proportion of participants |  | 0.2273 [0.0792 to 0.4208]

12. Secondary Outcome: Cumulative Incidence of Disease Relapse/Progression After Transplantation of Hematopoietic Cells Mobilized With BL-8040 (Arm 2 Recipients Only)
Description: -Disease relapse occurs in recipients who entered transplant in CR. Progression occurs in recipients with existent disease at transplant who meet criteria for progressive disease post-transplant. A recipient will be considered relapsed when there is a recurrence of the original malignant disease after transplantation. Date of relapse/progression is defined as the date at which the first observation of hematologic, radiographic, or cytogenetic changes which signify progression/relapse is made
Time Frame: At 1 year post-tranplantation
Population: Donors are not evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
proportion of participants |  | 0.227 [0.079 to 0.420]

13. Secondary Outcome: Cumulative Incidence of Disease Relapse/Progression After Transplantation of Hematopoietic Cells Mobilized With BL-8040 (Arm 2 Recipients Only)
Description: as for outcome 12
Time Frame: At 2 years post-tranplantation
Population: Donors are not evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
proportion of participants |  | 0.273 [0.107 to 0.470]

14. Secondary Outcome: Kaplan-Meier Estimate of Event Free Survival After Transplantation of Hematopoietic Cells Mobilized With BL-8040 (Arm 2 Recipients Only)
Description: -An event is defined as either graft failure, disease relapse as evidenced by hematologic, radiographic, or cytogenetic changes, or death. The event free survival is the time from Day 0 to occurrence of the first event.
Time Frame: At 2 years post-transplantation
Population: Donors are not evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
percentage of participants |  | 50.0

15. Secondary Outcome: Kaplan-Meier Estimate of Event Free Survival After Transplantation of Hematopoietic Cells Mobilized With BL-8040 (Arm 2 Recipients Only)
Description: as for outcome 14
Time Frame: At 3 years post-transplantation
Population: Donors are not evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
percentage of participants |  | 34.1

16. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival After Transplantation of Hematopoietic Cells Mobilized With BL-8040 (Arm 2 Recipients Only)
Description: -The time from Day 0 to death
Time Frame: At 2 years post-transplantation
Population: Donors are not evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
percentage of participants |  | 63.6

17. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival After Transplantation of Hematopoietic Cells Mobilized With BL-8040 (Arm 2 Recipients Only)
Description: -The time from Day 0 to death
Time Frame: At 3 years post-transplantation
Population: Donors are not evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 0 | 22
percentage of participants |  | 49.0

18. Secondary Outcome: Median Peripheral Blood CD34+ Cell Count (Arm 1 Donor Only)
Time Frame: At 3-4 hours after BL-8040
Population: Recipients are not evaluable for this outcome measure.
Measure: Median (Full Range); unit: CD34/microliters
Arm/Group | Arm 1: Donors | Arm 2: Recipients
Number analyzed (Participants) | 25 | 0
CD34/microliters | 15 [1 to 46] |

ADVERSE EVENTS:
Time Frame: -Adverse events for donors were collected from the date the participant signed the consent form through 30 days after the last dose of BL-8040. In addition, any adverse events at least possibly related to BL-8040 that occurs up to 5 years after the BL-8040 dose should be recorded. -Adverse events for recipients were collected from the start of the conditioning regimen until Day +100 post transplant. Only grade 3-5 non-hematologic adverse events will be collected.
Arm/Group | Arm 1: Donors | Arm 2: Recipients
All-Cause Mortality (participants affected / at risk) | 0/25 | 13/22
Serious Adverse Events (participants affected / at risk) | 0/25 | 12/22
Other Adverse Events (participants affected / at risk) | 25/25 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Donors (N=25) | Arm 2: Recipients (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 3
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Generalized weakness (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 3
Genital edema (Reproductive system and breast disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Donors (N=25) | Arm 2: Recipients (N=22)
Anemia (Blood and lymphatic system disorders) | 17 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 7
Acute systolic heart failure (Cardiac disorders) | 0 | 1
Chest pain-cardiac (Cardiac disorders) | 0 | 1
Sinus brachycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Eye pain (Eye disorders) | 1 | 0
Watering eyes (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 7
Nausea (Gastrointestinal disorders) | 5 | 2
Oral dysesthesia (Gastrointestinal disorders) | 6 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Edema limbs-anasarca (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 2
Fever (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 1 | 0
Injection site reaction (General disorders) | 20 | 0
Localized edema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Vibration sensation (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 20 | 0
Bacteremia-Klebsiella pneumoniae (Infections and infestations) | 0 | 1
Bacteremia-VRE (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Clostridium difficile (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 0 | 2
Oral thrush (Infections and infestations) | 0 | 1
Papulopustular rash (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
GGT increased (Investigations) | 0 | 1
Hemoglobin increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 7 | 0
Lymphocyte count increased (Investigations) | 22 | 0
Platelet count decreased (Investigations) | 22 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 2 | 0
A1c increased (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 10 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Foot pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Numbness in arms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysesthesia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 3
Paresthesia (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Scrotal pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 11 | 11
Hypotension (Vascular disorders) | 2 | 1
Veno-occlusive disease (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT02639559/Prot_SAP_000.pdf